CLINICAL TRIAL: NCT06803160
Title: Comparative Study of Laparoscopic Combined Trans-vesical and Extravesical Versus Laparoscopic Extravesical Fistula Excision in Uterovesical Fistula Repair: A Retrospective Observational Study
Status: Enrolling by invitation | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mahmoud Hossam, Mahmoud HossamEldin Saad Abdelhamid, Ain Shams University
Other Study IDs: Lap Uterovesical Fistula
Record Dates: First submitted 2025-01-26; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Success of Operation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Laparoscopic Combined Fistula Excision of Uterovesical Fistula: Patinets who underwent Laparoscopic Combined Fistula Excision of Uterovesical Fistula
  Interventions: Procedure: Laparoscopic Extravesical Fistula Excision of Uterovesical Fistula; Procedure: Laparoscopic Combined Fistula Excision of Uterovesical Fistula

INTERVENTIONS:
Procedure: Laparoscopic Extravesical Fistula Excision of Uterovesical Fistula — • In extravesical approach, the posterior bladder wall and the anterior uterine wall around the fistula will be dissected. Scar tissue around the orifice of the fistula will be removed and trimmed. After suturing uterine and bladder wall, intervening omentum will be placed in-between.
Procedure: Laparoscopic Combined Fistula Excision of Uterovesical Fistula — • In the combined approach, bladder will be opened bivalved till the site of the fistula. Scar tissue around the orifice of the fistula will be removed and trimmed. Careful dissection around the bladder and uterus will be done to suture both walls and place an intervening omentum in-between.

SUMMARY:
• The aim of this study is to compare between laparoscopic combined trans-vesical and extravesical versus laparoscopic extravesical fistula excision in uterovesical fistula repair.

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed with uterovesical fistula with history of uterine cesarean section or any urogenital surgery complaining of amenorrhea, cyclic hematuria, with or without urinary incontinence.

Exclusion Criteria:

* • Pregnant females.

  * Patients who refuse to participate in the study.
  * Patients with concomitant pathology that could affect symptoms e.g., polycystic ovary disease, stress incontinence, bladder cancer or overactive bladder.
  * Patients with malignant fistula.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: * This is a retrospective study involving the retrieval and analysis of medical records of uterovesical patients who were managed at the Urology and Gynecology departments at Ain Shams University Hospitals.
  * Patient's records that were included in the study satisfied the following criteria:
    * The patient was diagnosed with uterovesical fistula.
    * The patient had laparoscopic surgery with either approach at the Urology and Gynecology departments at Ain Shams University Hospitals.
    * The fistulous track was confirmed and had been repaired.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-01-30 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
success of operation | 6 months
  Success of operation with excision of fistula in upcoming CT cystogram

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol